CLINICAL TRIAL: NCT02020239
Title: The Effect of Physical Activity Intervention Flexibility on the Time Course of Changes in Body Composition and Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Cereal Partners Worldwide (Industry)
Responsible Party: Principal Investigator, Dr Andrew Blannin, Dr (PhD), Lecturer, University of Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bham_CPW_PhysActIntervention
Record Dates: First submitted 2013-12-12; First posted 2013-12-24 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Sedentary; Overweight
Keywords: physical activity; females; body composition
MeSH Terms: conditions — Sedentary Behavior; Overweight; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Prescribed exercise (Experimental): Participants will be asked to choose one activity and stick to it for the duration of the intervention. Participants will be able to choose between brisk walking/slow jogging or cycling. The intervention will require the completion of 30 minutes of chosen activity on 5 days of the week, which will be recorded in a physical activity diary.
  Interventions: Other: Exercise
- Points-based physical activity (Experimental): Participants will be asked to achieve a pre-set, individualised points target for physical activity each week. Points are acquired through the completion of a minimum 10 minutes of activity, choosing from the extensive list of activities provided; for example, 10 minutes of jogging achieves 4.5 points, whereas 10 minutes of washing a car achieves 1.5 points. The target will be 35-40 points per week, which equates to approximately 6 points per day. Any combination of activity, duration and frequency can be selected.
  Interventions: Other: Exercise
- Waiting list control (No Intervention): Participants will be asked to maintain their normal activities and diet. They will be added to a waiting list to receive either exercise intervention after completing the 24-week trial period, so that they do not miss out on the opportunity to receive the exercise intervention.

INTERVENTIONS:
Other: Exercise
  Arms: Points-based physical activity; Prescribed exercise

SUMMARY:
The investigators goal is to optimise physical activity interventions to help previously inactive women improve their body shape and composition. Many people seeking to lose weight or improve body composition initiate an exercise programme. The most common recommendation of an exercise intervention for someone attempting to manage their weight, has been to 'prescribe' the recommended 150 minutes of exercise per week (World Health Organisation), often using one mode of exercise. An alternative approach might be to offer a portfolio of activities, from which the exerciser can pick and choose, to facilitate greater amounts of physical activity. The problem with this is how do you account for the different intensities of walking, washing the car, playing badminton, cycling, jogging, etc? In this study, the investigators will try to overcome this barrier by allocating a number of "physical activity points" to each activity. Using this physical activity points system, participants will be provided with a points target that they can meet using any combination of activities.

The investigators research aim is therefore to compare this points-based system against the traditional 5x30minute prescription (and sedentary control) for their ability to help previously inactive women to drop a dress size, increase fat burning, positively change their body composition and tone their tummy.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 25-50 years old
* Inactive (less than 150 minutes of moderate-intensity aerobic physical activity per week)
* BMI 25-35 kg/m2
* Good general health, as assessed by the School of Sport, Exercise and Rehabilitation Sciences' General Health Questionnaire
* Willing to strictly comply with all study procedures and restrictions
* Willing to participate, as demonstrated by voluntary written informed consent

Exclusion Criteria:

* Positive result from the urine sample pregnancy test
* Currently breast feeding
* Currently participating in another clinical trial deemed to potentially interfere with this study
* Current or recent (within the last 30 days) smoker
* Currently taking prescription or non-prescription medication that may interfere with metabolism (including beta-blockers, insulin, bronchodilators, anti-inflammatory agents, thyroxine and medication/supplements that in the opinion of the investigators may affect metabolism).

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in body composition (fat and fat-free mass in kg) | 4 weeks, 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Perceived body shape | 4 weeks, 12 weeks and 24 weeks
Maximal aerobic capacity | 4 weeks, 12 weeks, 24 weeks
Fat oxidation rates | 4 weeks, 12 weeks and 24 weeks
Body tone | 4 weeks, 12 weeks, 24 weeks

OTHER OUTCOMES:
Blood-borne markers of metabolic health | 4 weeks, 12 weeks, 24 weeks
Psychological measures relating to perceived body image | 4 weeks, 12 weeks, 24 weeks
Psychological measures of attitudes towards exercise and physical activity | 4 weeks, 12 weeks, 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Birmingham, School of Sport, Exercise and Rehabilitation Sciences, Birmingham, United Kingdom

REFERENCES:
- [Derived] Holliday A, Burgin A, Fernandez EV, Fenton SAM, Thielecke F, Blannin AK. Points-based physical activity: a novel approach to facilitate changes in body composition in inactive women with overweight and obesity. BMC Public Health. 2018 Feb 17;18(1):261. doi: 10.1186/s12889-018-5125-2. PMID 29454318